CLINICAL TRIAL: NCT05785338
Title: Diagnosis of Fetal Isolated Cleft Palate Using Assessment of the Posterior Hard Palate Angle
Brief Title: Trial Observationnal
Acronym: CLEFTPALATDIAG
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Trial Observationnal
Record Dates: First submitted 2023-03-11; First posted 2023-03-27 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-03

CONDITIONS: Fetal Anomaly; Ultrasound
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- affected: patiente suspected for a cleft palate without cleft lip
  Interventions: Diagnostic Test: Posterior angle of the hard palate
- control: unaffected cases
  Interventions: Diagnostic Test: Posterior angle of the hard palate

INTERVENTIONS:
Diagnostic Test: Posterior angle of the hard palate — Fetal ultrasound
  Other Names: Gap within the hard palate and the no visualization of the nasal spine

SUMMARY:
The aim of this retrospective longitudinal study was to describe a key factor in the prenatal diagnosis of isolated cleft palate on the axial transverse view, in order to provide better understanding, detection and diagnosis of this anomaly.

DETAILED DESCRIPTION:
Objective: The study aims to evaluate the role of the posterior hard palate angle in the prenatal diagnosis of cleft palate.

Methods: Stored images of the axial transverse view of the fetal secondary palate, obtained at three-level ultrasounds, were used to evaluate the posterior border of the hard palate. The investigators studied the visualization of the posterior nasal spine and the presence of a gap within the hard palate. The investigators also assessed the posterior angle of the hard palate, formed by the posterior borders of the palatine bones next to the most posterior middle point of the palatine bone. The study population comprised 65 consecutive pregnancies of unaffected cases and 17 pregnancies with 24 assessments at different time points, suspected for a cleft palate without cleft lip, including 7 cases of cleft palate, 4 cases of high arched palate and 6 false positive cases.

ELIGIBILITY:
Inclusion Criteria:

- all patients suspected for a cleft palate without cleft lip referred to the Multidisciplinary Center for Prenatal Diagnosis in Poitiers (France) between January 2019 and January 2023.

Exclusion Criteria for the control group:

* major congenital anomalies or chromosomal aberration,
* premature rupture of the membranes,
* fetal demise,
* patients aged under 18 years.
* If the available images did not allow the evaluation of the hard palate, the case was excluded from further consideration.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnancy
Study Population: We included all patients suspected for a cleft palate without cleft lip (18 pregnant women with 24 assessments at different time points), referred to the Multidisciplinary Center for Prenatal Diagnosis in Poitiers (France) between January 2019 and January 2023. We compared the suspected group with 65 unaffected consecutive singleton pregnancies between 17 and 37 weeks, identified from our ultrasound database from June 2022 to Auguste 2022.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Rate of cleft palate without cleft lip | derivery
  Presence of cleft palate without cleft lip in postnatal exam

CONTACTS AND LOCATIONS:
Overall Officials: Iglika Simeonova-Brachot, MD, Principal Investigator — CHU Poitiers
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No